CLINICAL TRIAL: NCT01096719
Title: The Effect of Diets Targeting Energy Density and Energy Restriction on Weight Loss and Feelings of Deprivation, Satisfaction, and Hunger During Behavioral Weight Loss Treatment.
Brief Title: The Healthy Eating Choices for Life Program
Acronym: HEC4L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 8107 B
Record Dates: First submitted 2010-03-24; First posted 2010-03-31 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: Weight; Dietary intake; Energy Density; Behavioral; Satiety; Deprivation; Hunger; Fruit; Vegetable
MeSH Terms: conditions — Obesity; Body Weight; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Energy Density (Experimental)
  Interventions: Behavioral: Standard Behavioral Weight Loss Intervention; Behavioral: Dietary Goal: Reduction in Energy Density of Dietary Intake
- Lifestyle Treatment (Active Comparator)
  Interventions: Behavioral: Standard Behavioral Weight Loss Intervention; Behavioral: Dietary Goal: Reduction of Energy Intake
- Energy Density + Lifestyle Treatment (Experimental)
  Interventions: Behavioral: Standard Behavioral Weight Loss Intervention; Behavioral: Dietary Goal: Reduction in Energy Density of Dietary Intake; Behavioral: Dietary Goal: Reduction of Energy Intake

INTERVENTIONS:
Behavioral: Standard Behavioral Weight Loss Intervention — 12 week standard behavioral weight loss intervention including a physical activity goal and behavioral weight control strategies
Behavioral: Dietary Goal: Reduction in Energy Density of Dietary Intake — Consume low ED foods (ED < 1.0) for at least 10 items consumed per day and limit high ED foods (ED > 3.0) to two items consumed per day.
  Arms: Energy Density; Energy Density + Lifestyle Treatment
Behavioral: Dietary Goal: Reduction of Energy Intake — Limit energy intake to 1200 to 1500 kcals/day and < 30% kcals from fat.
  Arms: Energy Density + Lifestyle Treatment; Lifestyle Treatment

SUMMARY:
The purpose of this investigation is to conduct a 12-week pilot study to examine the effect of three different dietary prescriptions that differ on targeting reducing energy density (kcal/gram) and energy (kcal) on overall dietary intake, hunger, feelings of deprivation, satisfaction with the diet, mood, and weight loss in 45 overweight/obese adults receiving a 12-week behavioral weight loss intervention.

DETAILED DESCRIPTION:
Given the current prevalence of overweight and obesity among adults in the United States and the projected increase of these conditions in the future, development of effective weight loss and weight loss maintenance strategies is imperative. For weight loss to occur, energy intake needs to be reduced to incur an energy deficit, and for successful weight loss maintenance, energy intake needs to remain lower than energy intake at pre-weight loss levels due to an overall reduction in body size which reduces basal metabolic rate. One dietary strategy that may facilitate weight loss maintenance is consuming a diet low in dietary energy density (ED). This pilot study will test the effects of a dietary prescription focused on ED.

All participants in the investigation will receive a standard 12-week behavioral obesity intervention. The intervention will include an activity goal that participants will gradually work to achieve over the course of the 12-week intervention along with standard behavioral weight loss strategies. One condition will receive a dietary prescription for weight loss that focuses solely on lowering the ED of the diet, another condition will receive the traditional dietary prescription used in behavioral weight loss interventions that reduces energy intake, and the third condition will receive both prescriptions. Pre and post intervention measurements will be taken to determine if there are differences between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 65 years
* Body mass index (BMI) between 25 and 45 kg/m2

Exclusion Criteria:

* Report a health condition on the Physical Activity Readiness Questionnaire (PAR-Q)
* Report being unable to walk for 2 blocks (1/4 mile) without stopping
* Report major psychiatric diseases/organic brain syndromes via a phone screen
* Are currently participating in a weight loss program and/or taking weight loss medication or lost > 5% of body weight during the past 6 months
* Intend to move to another city within the time frame of the investigation
* Are pregnant, lactating, less than 6 months post-partum, or plan to become pregnant during the time frame of the investigation
* Have had gastric surgery for weight loss

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Energy density of the diet | Weeks 0 and 13
  Energy density is defined as the kilocalories per gram of a food. Energy density will be measured by collecting and analyzing 3-day food records using Nutrition Data Systems for Research at baseline (week 0) and post intervention (week 13).

SECONDARY OUTCOMES:
Weight Loss | Weeks 0 and 13
Feelings of dietary deprivation and satisfaction | Weeks 0 and 13
  Dietary deprivation and satisfaction will be measures using 100mm visual analog scales with the statements "I feel like I ate enough today" and "I feel like I ate what I wanted today". Both scales are anchored with "strongly disagree" on one end and "strongly agree" on the other end. These will be collected for 7 days at baseline (week 0) and post intervention (week 13).
Hunger | Weeks 0 and 13
  Hunger will be measured using a 100mm visual analog scale. The scale asks "How hungry did you feel today?" and is anchored with "not at all hungry" on one end and "extremely hungry" on the other. Hunger scales will be collected for 7 days at baseline (week 0) and post intervention (week 13).

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, RD, LDN, Principal Investigator — University of Tennessee
Locations (1):
- Healthy Eating and Activity Laboratory, Knoxville, Tennessee, United States

REFERENCES:
- [Derived] Raynor HA, Steeves EA, Hecht J, Fava JL, Wing RR. Limiting variety in non-nutrient-dense, energy-dense foods during a lifestyle intervention: a randomized controlled trial. Am J Clin Nutr. 2012 Jun;95(6):1305-14. doi: 10.3945/ajcn.111.031153. Epub 2012 May 2. PMID 22552025
- See also: Healthy Eating and Activity Laboratory Homepage — http://heal.utk.edu/